CLINICAL TRIAL: NCT05165329
Title: A Randomised, Controlled Trial Evaluating the Effectiveness of Probiotic and Peanut Oral Immunotherapy (PPOIT) in Inducing Desensitisation or Remission in Chinese Children With Peanut Allergy Compared With Oral Immunotherapy (OIT) Alone and With Placebo
Brief Title: A Randomized, Controlled Trial of Probiotic and Peanut Oral Immunotherapy (PPOIT) in Inducing Tolerance in Hong Kong Children With Peanut Allergy Compared With Oral Immunotherapy (OIT) Alone and With Placebo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ting-fan Leung, Professor Ting-fan Leung, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPOIT-HK
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Peanut Allergy; Food Allergy in Children
Keywords: peanut allergy; oral immunotherapy; sustained unresponsiveness; tolerance
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Food Coloring Agents; Taste

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic and Peanut Oral Immunotherapy (PPOIT) (Active Comparator): Probiotic and peanut oral immunotherapy taken daily for 18 months
  Interventions: Combination Product: PEANUT OIT: Peanut Flour (50% peanut protein) that is prepared under food manufacturing regulations
- Placebo Probiotic and Peanut Oral Immunotherapy (Active Comparator): Placebo probiotic and peanut oral immunotherapy taken daily for 18 months
  Interventions: Combination Product: PEANUT OIT: Peanut Flour (50% peanut protein) that is prepared under food manufacturing regulations
- Placebo Probiotic and Placebo Oral Immunotherapy (Placebo Comparator): Placebo probiotic and placebo oral immunotherapy taken daily for 18 months
  Interventions: Combination Product: PEANUT PLACEBO: Peanut Placebo is maltodextrin powder with food colouring and peanut essence that has similar appearance, taste and smell to the active product.

INTERVENTIONS:
Combination Product: PEANUT OIT: Peanut Flour (50% peanut protein) that is prepared under food manufacturing regulations — PROBIOTIC: The probiotic to be used is Lactobacillus rhamnosus GG, supplied as a freeze-dried powder. Probiotic will be prepared under strict Food Manufacturing Regulations. The daily dose of 2x10^10 cfu will be packed individually in sachets. Participants will be instructed to mix one scoop of the probiotic in water at a temperature NOT exceeding 38 degrees Celsius. The probiotic must be stored at 4 degrees Celsius
  Arms: Probiotic and Peanut Oral Immunotherapy (PPOIT)
Combination Product: PEANUT OIT: Peanut Flour (50% peanut protein) that is prepared under food manufacturing regulations — PROBIOTIC PLACEBO: Probiotic Placebo is maltodextrin. The daily dose will be measured using a standardised scoop. Participants will be instructed to mix one scoop of the probiotic in water at a temperature NOT exceeding 38 degrees Celsius. The probiotic should be stored at 2-8 degrees Celsius.
  Arms: Placebo Probiotic and Peanut Oral Immunotherapy
Combination Product: PEANUT PLACEBO: Peanut Placebo is maltodextrin powder with food colouring and peanut essence that has similar appearance, taste and smell to the active product. — PROBIOTIC PLACEBO: Probiotic Placebo is maltodextrin. The daily dose will be measured using a standardised scoop. Participants will be instructed to mix one scoop of the probiotic in water at a temperature NOT exceeding 38 degrees Celsius. The probiotic should be stored at 2-8 degrees Celsius.
  Arms: Placebo Probiotic and Placebo Oral Immunotherapy

SUMMARY:
At present there is no cure for food allergy. People with a food allergy need to avoid the food they are allergic to in order to stay safe. However we know that accidental exposure is common. Researchers have begun to look at the effectiveness of 'oral immunotherapy' as a treatment for food allergy but results have been mixed.

This study is a randomized controlled trial to evaluate the effectiveness of Probiotic and Peanut Oral Immunotherapy (PPOIT) in inducing tolerance in children with peanut allergy compared with Oral Immunotherapy (OIT) alone and with Placebo. Children will take increasing doses of peanut protein and a set amount of probiotic until a total of 18 months treatment is completed. Children will be tested for peanut allergy at the start of the study, at the end of PPOIT treatment T1 (18 months) and T2 (8 weeks) and T3 (1year) after treatment.

DETAILED DESCRIPTION:
This is a three-armed, randomised (4:4:1), stratified (by age), blinded, placebo-controlled, parallel-group, superiority trial.

1. PPOIT Probiotic and peanut OIT taken daily for 18 months.
2. OIT Probiotic placebo and peanut OIT taken daily for 18 months.
3. Placebo Probiotic placebo and OIT placebo taken daily for 18 months.

The study consists of:

Screening visit occurs within three months before Day 1.

Day 1 Rush Induction Phase is the start of treatment where participants receive increasing doses of peanut (or placebo) OIT every 20 minutes to reach a final dose of 12mg of peanut protein (or placebo). A single dose of 2x10^10 cfu Lactobacillus rhamnosus GG (or placebo) is also taken.

Week 1 - 16 is the Buildup Phase where the daily dose of peanut (or placebo) OIT is increased every 2 weeks* until a maintenance dose of 2000mg peanut protein (or placebo) is reached. This is expected to take 16 weeks. A fixed daily dose of 2x10^10 cfu Lactobacillus rhamnosus GG (or placebo) is taken during this phase.

* In unavoidable circumstances i.e. school camps, examinations, when scheduling must be amended depending on parents/ participants availability, the window for buildup visits can be +/- 7 days.

Week 16 - 78 is the Maintenance Phase where participants take a daily dose of 2g of peanut protein (or placebo) and a daily dose of 2x10^10 cfu Lactobacillus rhamnosus GG (or placebo) at home and continue until a total of 18 months of treatment is completed.

Week 78 - 86 is the Elimination Phase where participants continue on a peanut-elimination diet post-treatment.

Week 86 -130 is the Monitoring Phase: All groups will be followed up for 12 months after the treatment period. During this time, at 6 months, a telephone interview will be conducted with the participant's parent or guardian to collect information on exposure to peanut/amount of peanut being eaten and allergic reactions.

The primary outcome analysis will be conducted when all subjects have either completed the T2 DBPCFC or terminated the study prior to their T2 visit. Analysis of safety and tolerability, and other secondary outcomes to the T2 timepoint will also be conducted at this time. A supplemental analysis will be conducted at the end of study (i.e. when last subject completes T3 or has withdrawn from the study prior to their T3 visit, or sponsor terminates the study), using cumulative data from the study.

ELIGIBILITY:
Inclusion Criteria: Subjects are eligible if they meet all of the following criteria

* Aged between 1 year and 17 years of age;
* >=7kg (the weight considered safe for administration of adrenaline autoinjector (e.g. Jext);
* Ethnic Chinese; and
* Confirmed diagnosis of peanut allergy as defined by a failed double-blind placebo-controlled food challenge (DBPCFC) with peanut and a serum peanut-specific IgE level of at least 0.35 kUA (allergen-specific unit) per liter according to ImmunoCAP (Thermo Fisher Scientific) at screening.

Exclusion Criteria: Subjects are not eligible if they meet any of the following criteria

* History of severe anaphylaxis (as defined by persistent hypotension, collapse, loss of consciousness, persistent hypoxia or ever needing >3 doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction);
* Severe anaphylaxis during the study entry DBPCFC (defined as persistent hypotension, collapse, loss of consciousness, persistent hypoxia, or requiring >3 doses of intramuscular adrenaline or an intravenous adrenaline infusion for management of an allergic reaction);
* FEV1 <85% at rest and FEV1/FVC ≤ 85% at rest or ongoing chronic persistent asthma (as per Australian Asthma Foundation guidelines);
* Underlying medical conditions (e.g. cardiac disease) that increase the risks for anaphylaxis;
* Use of beta-blockers, and ACE inhibitors;
* Inflammatory intestinal conditions, indwelling catheters, gastrostomies, immunocompromised states, post-cardiac and/or gastrointestinal tract surgery, critically-ill or other conditions that may increase the risks of probiotic associated sepsis;
* Already taking probiotic supplements or foods containing probiotics within the past month;
* Reacting to the placebo component during the study entry DBPCFC;
* Have received other food immunotherapy treatment in the preceding 12 months;
* History of suspected or biopsy-confirmed eosinophilic esophagitis (EoE);
* Currently taking immunomodulatory therapy (including allergen immunotherapy);
* Past or current major illness that in the opinion of the Site Investigator may affect the subject's ability to participate in the study e.g. increased risk to the participant;
* Subjects who in the opinion of the Site Investigator are unable to follow the protocol;
* Another family member already enrolled in the trial (to maintain safety and blinding); or
* Non-English and non-Chinese speaking participants and their families. NOTE: participants with other food allergies are NOT excluded from participating in this trial.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with 8-week sustained unresponsiveness (passed T1 and T2 challenges) in PPOIT vs placebo | T2 - 8 weeks after final day of maintenance treatment

SECONDARY OUTCOMES:
Proportion of participants with 8-week sustained unresponsiveness (passed T1 and T2 challenges) in PPOIT vs peanut OIT. | T2 - 8 weeks after final day of maintenance treatment
Proportion of participants who achieve full desensitisation (passed T1 challenge) in: (i) PPOIT vs placebo and (ii) PPOIT vs OIT; and (iii) OIT vs placebo. | T1 - One Day after final day of maintenance treatment
The cumulative dose tolerated during the T1 challenge in: (i) PPOIT vs placebo and (ii) PPOIT vs OIT; and (iii) OIT vs placebo. | T1 - One Day after final day of maintenance treatment
  Cumulative doses below the reaction-eliciting dose if there is a reaction; or total cumulative challenge dose if there is no reaction
Peanut SPT wheal size and peanut and peanut component (Ara h 1, Ara h 2, Ara h 3) sIgE and sIgG4 levels in: (i) PPOIT vs placebo; (ii) PPOIT vs OIT; and (iii) OIT vs placebo and their correlation with sustained unresponsiveness. | At 12 months of treatment; T1 - One Day after final day of maintenance treatment. T2 - 8 weeks after final day of maintenance treatment
Exposure-adjusted incidence rate and severity of treatment emergent adverse events (TEAEs) in (i) PPOIT vs placebo; and (ii) PPOIT vs OIT; and (iii) OIT vs placebo groups. | TEAEs will be collected until T2 - 8 weeks after final day of maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Fan Leung, Principal Investigator — Chinese University of Hong Kong
Locations (4):
- Hong Kong (4):
  - Department of Paediatrics and Adolescent Medicine, Hong Kong Children's Hospital, Hong Kong
  - Department of Paediatrics and Adolescent Medicine, Princess Margaret Hospital, Hong Kong
  - Department of Paediatrics, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong
  - Department of Paediatrics, Queen Elizabeth Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.allergycuhk.org/ppoit-hk